CLINICAL TRIAL: NCT00475865
Title: A Randomized, Multinational, Double-blind, Placebo-controlled, Parallel-group Design Pilot Study to Estimate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamic Effects of Teriflunomide for 24 Weeks When Added to Treatment With Glatiramer Acetate in Subjects With Multiple Sclerosis
Brief Title: Phase II Study of Teriflunomide as Adjunctive Therapy to Glatiramer Acetate in Subjects With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDY6046; 2006-004893-29 (EudraCT Number); HMR1726D-2004 (Other: HMR)
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Results first posted 2012-11-02 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: MS; glatiramer acetate; adjunctive therapy; relapses
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — teriflunomide; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + GA (Placebo Comparator): Placebo (for teriflunomide) once daily concomitantly with glatiramer acetate (GA) for 24 weeks
  Interventions: Drug: Placebo (for teriflunomide); Drug: Glatiramer Acetate (GA)
- Teriflunomide 7 mg + GA (Experimental): Teriflunomide 7 mg once daily concomitantly with glatiramer acetate (GA) for 24 weeks
  Interventions: Drug: Teriflunomide; Drug: Glatiramer Acetate (GA)
- Teriflunomide 14 mg + GA (Experimental): Teriflunomide 14 mg once daily concomitantly with glatiramer acetate (GA) for 24 weeks
  Interventions: Drug: Teriflunomide; Drug: Glatiramer Acetate (GA)

INTERVENTIONS:
Drug: Teriflunomide — Film-coated tablet
  Oral administration
  Other Names: HMR1726
  Arms: Teriflunomide 14 mg + GA; Teriflunomide 7 mg + GA
Drug: Placebo (for teriflunomide) — Film-coated tablet
  Oral administration
  Arms: Placebo + GA
Drug: Glatiramer Acetate (GA) — Solution in prefilled syringe for subcutaneous injection
  Other Names: Copaxone®

SUMMARY:
The primary objective was to estimate the tolerability and safety of 2 doses of Teriflunomide administered once daily for 24 weeks, compared to placebo, in patients with multiple sclerosis [MS] with relapses who were on a stable dose of Glatiramer Acetate [GA].

The secondary objectives were:

* to estimate the effect of the 2 doses of Teriflunomide, compared to placebo, in combination with a stable dose of GA on Magnetic Resonance Imaging [MRI] parameters, relapse rate and patient-reported fatigue;
* to perform pharmacokinetic analyses of the 2 doses of teriflunomide in combination with a stable dose of GA.

DETAILED DESCRIPTION:
The duration of the study period for a participant was approximatively 44 weeks broken down as follows:

* Screening period up to 4 weeks,
* 24-week double-blind treatment period*,
* 16-week post-treatment elimination follow-up period.

'*' Participants successfully completing the week 24 visit were offered the opportunity to enter the optional long-term extension study LTS6047 - NCT00811395.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to McDonald's criteria;
* Relapsing clinical course, with or without progression;
* Expanded Disability Status Scale [EDSS] less or equal to 5.5 (ambulatory);
* Stable dose of Glatiramer Acetate [GA] for at least 26 weeks prior to the screening visit;
* No onset of MS relapse in the preceding 60 days prior to randomization;
* Clinically stable for 4 weeks prior to randomization.

Exclusion Criteria:

* Other chronic disease of the immune system, liver function impairment or chronic pancreatic disease;
* Pregnant or nursing woman;
* Alcohol or drug abuse;
* Use of cladribine, Mitoxantrone, or other immunosuppressant agents such as Azathioprine, Cyclophosphamide, Cyclosporin, Methotrexate or Mycophenolate before enrollment;
* Human immunodeficiency virus [HIV] positive status;
* Any known condition or circumstance that would prevent in the investigator's opinion compliance or completion of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (6):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Derived] Freedman MS, Wolinsky JS, Truffinet P, Comi G, Kappos L, Miller AE, Olsson TP, Benamor M, Chambers S, O'Connor PW. A randomized trial of teriflunomide added to glatiramer acetate in relapsing multiple sclerosis. Mult Scler J Exp Transl Clin. 2015 Dec 7;1:2055217315618687. doi: 10.1177/2055217315618687. eCollection 2015 Jan-Dec. PMID 28607708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment initiated in April 2007 was completed in December 2008.
  A total of 148 patients were screened at 24 sites in 6 countries.
Pre-assignment Details: Randomization was stratified by country.
  Assignment to groups was done centrally using an Interactive Voice Response System (IVRS] in a 1:1:1 ratio after confirmation of the selection criteria.
  123 participants were randomized.
Groups:
- Placebo + GA: Placebo (for teriflunomide) once daily concomitantly with Glatiramer Acetate [GA] for 24 weeks
- Teriflunomide 7 mg + GA: Teriflunomide 7 mg once daily concomitantly with Glatiramer Acetate [GA] for 24 weeks
- Teriflunomide 14 mg + GA: Teriflunomide 14 mg once daily concomitantly with Glatiramer Acetate [GA] for 24 weeks
Period: Overall Study
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Started | 41 (randomized) | 42 (randomized) | 40 (randomized)
Treated | 41 (completed treatment period) | 42 | 40
Completed | 39 | 37 (completed treatment period) | 34 (completed treatment period)
Not Completed | 2 | 5 | 6
Not completed — Adverse Event | 0 | 3 | 4
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 2
Not completed — Participant did not wish to continue | 1 | 0 | 0
Not completed — Other than above | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA | Total
Number analyzed (Participants) | 41 | 42 | 40 | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (8.5) | 42.1 (7.8) | 40.3 (7.5) | 41.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 32 | 97
  Male | 9 | 9 | 8 | 26
Region of Enrollment [Number; unit: participants] — Europe: Austria, Germany, Italy and United Kingdom
  North America: Canada and United States
  participants
    Europe | 23 | 22 | 21 | 66
    North America | 18 | 20 | 19 | 57
Time since first diagnosis of Multiple Sclerosis [MS] [Mean (Standard Deviation); unit: years] | 7.61 (6.04) | 8.82 (5.85) | 7.60 (6.03) | 8.02 (5.95)
Number of MS relapses [Median (Full Range); unit: MS relapses]
  Within the past year | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 4] | 1 [0 to 4]
  Within the past 2 years | 1 [0 to 5] | 1 [0 to 7] | 1 [0 to 6] | 1 [0 to 7]
Time since most recent MS relapse onset [Mean (Standard Deviation); unit: months] | 24.90 (34.84) | 21.52 (30.48) | 23.88 (31.53) | 23.41 (32.09)
MS subtype [Number; unit: participants]
  Relapsing Remitting | 39 | 40 | 37 | 116
  Secondary Progressive | 2 | 2 | 3 | 7
  Progressive Relapsing | 0 | 0 | 0 | 0
Baseline Expanded Disability Status Scale [EDSS] score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that qualifies disability in patients with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation.
  EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
  units on a scale | 2.54 (1.11) | 2.43 (1.23) | 2.60 (1.28) | 2.52 (1.20)

OUTCOME MEASURES:

1. Primary Outcome: Overview of Adverse Events (AE]
Description: AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: from first study drug intake up to 112 days after last intake or up to the first intake in the extension study LTS6047, whichever occured first (40 weeks max)
Population: All randomized and treated participants; Participants were included in the treatment group according to the drug actually received.
Measure: Number; unit: participants
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
participants
  Any AE | 32 | 35 | 35
  - serious AE | 3 | 3 | 1
  - AE leading to death | 0 | 0 | 0
  - AE leading to study drug discontinuation | 0 | 3 | 4

2. Primary Outcome: Overview of AE With Potential Risk of Occurrence
Description: AE with potential risk of occurrence were defined as follows:
  * Hepatic disorders;
  * Immune effects, mainly effects on bone marrow and infection;
  * Pancreatic disorders;
  * Malignancy;
  * Skin disorders, mainly hair loss and hair thinning;
  * Pulmonary disorders;
  * Hypertension;
  * Peripheral neuropathy;
  * Psychiatric disorders;
  * Hypersensitivity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
participants
  Any AE with potential risk of occurence | 24 | 28 | 28
  - Hepatic disorder AE | 4 | 2 | 5
  - Pancreatic disorder AE | 6 | 5 | 6
  - Pulmonary disorder AE | 0 | 1 | 0
  - Immune effects related AE | 18 | 18 | 15
  - Hair loss / Hair thinning AE | 1 | 5 | 7
  - Hypertension-related AE | 0 | 1 | 0
  - Peripheral neuropathy AE | 2 | 1 | 5
  - Hypersensitivity AE | 3 | 3 | 8
  - Malignancy AE | 0 | 0 | 0
  - Psychiatric disorder AE | 1 | 3 | 1

3. Primary Outcome: Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA)
Description: PCSA values are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review.
  Hepatic parameters thresholds were defined as follows:
  * Alanine Aminotransferase [ALT] >3, 5, 10 or 20 Upper Normal Limit [ULN];
  * Aspartate aminotransferase [AST] >3, 5, 10 or 20 ULN;
  * Alkaline Phosphatase >1.5 ULN;
  * Total Bilirubin [TB] >1.5 or 2 ULN;
  * ALT >3 ULN and TB >2 ULN.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
participants
  ALT >3 ULN | 1 | 0 | 1
  - ALT >5 ULN | 1 | 0 | 1
  - ALT >10 ULN | 1 | 0 | 0
  AST >3 ULN | 1 | 0 | 0
  - AST >5 ULN | 1 | 0 | 0
  Alkaline Phosphatase >1.5 ULN | 0 | 0 | 0
  TB >1.5 ULN | 0 | 0 | 0
  ALT >3 ULN and TB >2 ULN | 0 | 0 | 0

4. Secondary Outcome: Cerebral Magnetic Resonance Imaging [MRI] Assessment: Change From Baseline in Total Lesion Volume (Burden of Disease)
Description: Total lesion volume is the sum of the total volume of all T2-lesions and the total volume all T1-hypointense post-gadolinium lesions measured through T2/proton density scan analysis and gadolinium-enhanced T1 scan analysis.
  Least-square means were estimated using a Mixed-effect model with repeated measures [MMRM] on cubic root transformed volume data (treatment group, region of enrollment, visit, treatment-by-visit interaction, baseline value (cubic root transformed), and baseline-by-visit interaction as factors).
Time Frame: baseline (before randomization) and 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mililiters (mL)
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
mililiters (mL) | -0.006 (0.036) | -0.030 (0.036) | -0.036 (0.037)

5. Secondary Outcome: Cerebral MRI Assessment: Number of Gd-enhancing T1-lesions Per Scan (Poisson Regression Estimates)
Description: Number of Gd-enhancing T1-lesions per scan is obtained from the total number of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
  To account for the different number of scans among participants, a Poisson regression model with robust error variance was used (total number of Gd-enhancing T1-lesions as response variable; log-transformed number of scans as "offset" variable; treatment group, region of enrollment and baseline number of Gd-enhancing T1-lesions as covariates).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
lesions per scan | 0.367 [0.183 to 0.736] | 0.109 [0.054 to 0.220] | 0.171 [0.093 to 0.313]

6. Secondary Outcome: Cerebral MRI Assessment: Volume of Gd-enhancing T1-lesions Per Scan
Description: Total volume of Gd-enhancing T1-lesions per scan is obtained from the sum of the volumes of Gd-enhancing T1-lesions observed during the study divided by the total number of scans performed during the study.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: mililiters per scan
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
mililiters per scan | 0.063 | 0.028 | 0.017

7. Secondary Outcome: Annualized Relapse Rate [ARR]: Poisson Regression Estimates
Description: ARR is obtained from the total number of confirmed relapses that occured during the treatment period divided by the sum of the treatment durations.
  Each episode of relapse - appearance, or worsening of a clinical symptom that was stable for at least 30 days, that persisted for a minimum of 24 hours in the absence of fever - was to be confirmed by an increase in Expanded Disability Status Scale [EDSS] score or Functional System scores.
  To account for the different treatment durations among participants, a Poisson regression model with robust error variance was used (total number of confirmed relapses as response variable; log-transformed treatment duration as "offset" variable; treatment group and region of enrollment as covariates).
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 41 | 42 | 40
relapses per year | 0.475 [0.260 to 0.867] | 0.311 [0.151 to 0.642] | 0.647 [0.379 to 1.103]

8. Secondary Outcome: Pharmacokinetic [PK]: Teriflunomide Plasma Concentration
Description: Plasma concentrations of teriflunomide were measured using validated liquid chromatography-tandem mass spectrometry methods.
Time Frame: 24 weeks
Population: All randomized and treated participants who had at least one PK sample. Participants were included in the treatment group according to the drug actually received.
Measure: Mean (Standard Deviation); unit: micrograms/mililiter (μg/mL)
Arm/Group | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Number analyzed (Participants) | 37 | 33
micrograms/mililiter (μg/mL) | 23.443 (10.917) | 46.992 (32.154)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent Form up to the last visit.
Description: The analysis was performed on the exposed population and included all AE that developed or worsened from first study drug intake up to 112 days after last study drug intake or up to the first study drug intake in the extension study LTS6047, whichever occured first (40 weeks max)
Arm/Group | Placebo + GA | Teriflunomide 7 mg + GA | Teriflunomide 14 mg + GA
Serious Adverse Events (participants affected / at risk) | 3/41 | 3/42 | 1/40
Other Adverse Events (participants affected / at risk) | 20/41 | 20/42 | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + GA (N=41) | Teriflunomide 7 mg + GA (N=42) | Teriflunomide 14 mg + GA (N=40)
Abscess (Infections and infestations) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + GA (N=41) | Teriflunomide 7 mg + GA (N=42) | Teriflunomide 14 mg + GA (N=40)
Gastroenteritis (Infections and infestations) | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 4 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 5 | 6 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 8
Nausea (Gastrointestinal disorders) | 2 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 5
Fatigue (General disorders) | 6 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results of the work performed pursuant to this protocol. Prior to publication, the investigator provides the sponsor with the manuscript for review and comment at least 45 days in advance of its submission for publication.

The sponsor can require the investigator to withhold publication an additional 90 days to allow for filing a patent application or taking such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.